CLINICAL TRIAL: NCT00027274
Title: Etiologic Investigation of Cancer Susceptibility in Inherited Bone Marrow Failure Syndromes: A Natural History Study
Brief Title: Cancer in Inherited Bone Marrow Failure Syndromes
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020052; 02-C-0052; NCT00056121 (obsolete NCT alias)
Record Dates: First submitted 2001-11-29; First posted 2001-11-30 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Diamond Blackfan Anemia; Dyskeratosis Congenita; Fanconi Anemia; Shwachman Diamond Syndrome; Inherited Bone Marrow Failure Syndrome, Aplastic Anemia
Keywords: Fanconi Anemia; Diamond Blackfan Anemia; Dyskeratosis Congenita; Shwachman Diamond Syndrome; Hereditary; Natural History; Fanconi's Anemia; Bone Marrow; Inherited Bone Marrow Failure Syndromes; IBMFS; Familial Cancer
MeSH Terms: conditions — Anemia, Diamond-Blackfan; Dyskeratosis Congenita; Fanconi Anemia; Shwachman-Diamond Syndrome; Congenital Bone Marrow Failure Syndromes; Anemia, Aplastic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: All families with a member who has one of the relevant syndromes.

SUMMARY:
Background:

A prospective cohort of Inherited Bone Marrow Failure Syndrome (IBMFS) will provide new information regarding cancer rates and types in these disorders.

Pathogenic variant(s) in IBMFS genes are relevant to carcinogenesis in sporadic cancers.

Patients with IBMFS who develop cancer differ in their genetic and/or environmental features from patients with IBMFS who do not develop cancer.

These cancer-prone families are well suited for cancer screening and prevention trials targeting those at increased genetic risk of cancer.

Carriers of IBMFS pathogenic variant(s) are at increased risk of cancer.

The prototype disorder is Fanconi's Anemia (FA); other IBMFS will also be studied.

Objectives:

To determine the types and incidence of specific cancers in patients with an IBMFS.

To investigate the relevance of IBMFS pathogenic variant(s) in the carcinogenesis pathway of the sporadic counterparts of IBMFS-associated cancers.

To identify risk factors for IBMFS-related cancers in addition to the primary germline pathogenic variant(s).

To determine the risk of cancer in IBMFS carriers.

Eligibility:

North American families with a proband with an IBMFS.

IBMFS suspected by phenotype, confirmed by pathogenic variant(s) in an IBMFS gene, or by clinical diagnostic test.

Fanconi's anemia: birth defects, marrow failure, early onset malignancy; positive chromosome breakage result.

Diamond-Blackfan anemia: pure red cell aplasia; elevated red cell adenosine deaminase.

Dyskeratosis congenita: dysplastic nails, lacey pigmentation, leukoplakia; marrow failure.

Shwachman-Diamond Syndrome: malabsorption; neutropenia.

Amegakaryocytic thrombocytopenia: early onset thrombocytopenia.

Thrombocytopenia absent radii: absent radii; early onset thrombocytopenia.

Severe Congenital Neutropenia: neutropenia, pyogenic infections, bone marrow maturation arrest.

Pearson's Syndrome: malabsorption, neutropenia, marrow failure, metabolic acidosis; ringed sideroblasts.

Other bone marrow failure syndromes: e.g. Revesz Syndrome, WT, IVIC, radio-ulnar synostosis, ataxia-pancytopenia.

First degree relatives of IBMFS-affected subjects as defined here, i.e. siblings (half or full), biologic parents, and children.

Grandparents of IBMFS-affected subjects.

Patients in the general population with sporadic tumors of the types seen in the IBMFS (head and neck, gastrointestinal, and anogenital cancer), with none of the usual risk factors (e.g. smoking, drinking, HPV).

Design:

Natural history study, with questionnaires, clinical evaluations, clinical and research laboratory test, review of medical records, cancer surveillance.

Primary endpoints are all cancers, solid tumors, and cancers specific to each type of IBMFS.

Secondary endpoints are markers of pre-malignant conditions, such as leukoplakia, serum or tissue evidence of carcinogenic viruses, and bone marrow morphologic myelodyplastic syndrome or cytogenetic clones.

DETAILED DESCRIPTION:
Study Description:

This is a natural history study involving questionnaires, clinical and research evaluations, clinical and research laboratory tests, review of medical records, cancer surveillance. A prospective cohort of Inherited Bone Marrow Failure Syndrome (IBMFS) will provide new information regarding cancer rates and types in these disorders.

Pathogenic variant(s) in IBMFS genes are relevant to carcinogenesis in sporadic cancers.

This study will determine whether patients with IBMFS who develop cancer differ in their genetic and/or environmental features from patients with IBMFS who do not develop cancer.

These cancer-prone families are well suited for cancer screening and prevention trials targeting those at increased genetic risk of cancer.

Carriers of IBMFS gene pathogenic variant(s) are at increased risk of cancer.

The prototype disorder is Fanconi Anemia (FA); other IBMFS will also be studied.

Objectives:

To determine the types and incidence of specific cancers in patients with an IBMFS.

To investigate the relevance of IBMFS gene pathogenic variants in the carcinogenesis pathway of the sporadic counterparts of IBMFS-associated cancers.

To identify risk factors for IBMFS-related cancers in addition to the primary germline pathogenic variant(s).

To determine the risk of cancer in IBMFS carriers.

Endpoints:

Primary Endpoint:

-All cancers, solid tumors, and cancers specific to each type of IBMFS.

Secondary Endpints:

-Secondary endpoints are markers of pre-malignant conditions, such as leukoplakia, serum or tissue evidence of carcinogenic viruses, and bone marrow morphologic myelodyplastic syndrome or cytogenetic clones.

ELIGIBILITY:
* INCLUSION CRITERIA:

The participants will be affected by an IBMFS, or be members of a family with an IBMFS, and be at risk of being affected or carriers of the syndrome. Except for the rare X-linked recessive disorder (e.g. some dyskeratosis congenita patients), there should be equal numbers of male and female probands and family members. These IBMFS have been reported in most racial and ethnic groups, and thus all such groups will be included. The age range will be from birth to old age (grandparents of probands). The majority of the probands will be children (10-20% will be adults), and their parents and grandparents will be adults. All racial/ethnic groups are eligible.

INCLUSION CRITERIA for Patients:

* Fanconi s anemia.
* Diamond Blackfan anemia.
* Dyskeratosis congenita.
* Shwachman Diamond Syndrome.
* Amegakaryocytic thrombocytopenia.
* Thrombocytopenia absent radii.
* Severe Congenital Neutropenia.
* Pearson Syndrome.
* Other bone marrow failure syndromes.

Family Members of IBMFS - Affected Subjects:

-Family members include first degree relatives of IBMFS-affected subjects as defined here, i.e. siblings (half or full), biologic parents, and children. Grandparents of IBMFS-affected subjects are also included, specifically for Hypothesis 4. The age range will be from birth to old age (grandparents of probands).

Patients in the general population:

-Patients in the general population with sporadic tumors of the types seen in the IBMFS (head and neck, gastrointestinal, and anogenital cancer), with none of the usual risk factors for those tumors (e.g. smoking, drinking, HPV). These patients will be further evaluated for an IBMFS by the referring physician under the guidance of the study investigators and if diagnosed with an IBMFS or if not diagnosed but highly suspicious for an IBMFS, would be eligible for inclusion in the Field and Clinic Center cohorts.

EXCLUSION CRITERIA:

-Affected: An individual who meets any of the following criteria will be excluded from participation in this study:

* Evidence that the hematologic disorder is acquired rather than genetic. Such evidence includes temporal relation of the aplastic anemia to known marrow suppressant drugs, chemicals, toxins, or viruses (in the absence of evidence indicative of an inherited marrow failure disorder).
* Known causes of cytopenias such as autoantibodies to red cells, platelets, or neutrophils, viruses (especially hepatitis), micronutrient deficiencies, transient erythroblastopenia of childhood, and cyclic neutropenia.
* Assignment of the patient s physical findings to other syndromes or causes that are not part of the IBMFS disease spectrum.
* Inability of the participant or LAR to understand and be willing to sign a written informed consent document.
* Unwillingness to permit access to medical records and pathology specimens.

There are no other exclusion parameters not related to the primary disease.

-Unaffected/Family Members: An individual who meets any of the following criteria will be excluded from participation in this study:

* If there is no affected individual in the family who meets the inclusion criteria
* Inability of the participant or LAR to understand and be willing to sign a written informed consent document.
* Unwillingness to permit access to medical records and pathology specimens.

Ages: 1 Day to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All families with a member who has one of the relevant syndromes.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2001-11-28 (Actual)

PRIMARY OUTCOMES:
Cohort of Families with IBMFS | Ongoing
  Establish a cohort of families with IBMFS
Biology of Patients Compared with Healthy Controls | Ongoing
  Compare biology of IBMFS patients with general populations
Differences Between Patients and Healthy Controls | Ongoing
  Identify differences between patients with IBMFS who develop cancer and those who don't
Risk of Cancer with Specific Mutations | Ongoing
  Determine risk of cancer in IBMFS patients with specific gene mutations

CONTACTS AND LOCATIONS:
Overall Officials: Lisa J McReynolds, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - National Cancer Institute - Shady Grove, Rockville, Maryland

REFERENCES:
- [Background] Vlachos A, Rosenberg PS, Atsidaftos E, Alter BP, Lipton JM. Incidence of neoplasia in Diamond Blackfan anemia: a report from the Diamond Blackfan Anemia Registry. Blood. 2012 Apr 19;119(16):3815-9. doi: 10.1182/blood-2011-08-375972. Epub 2012 Feb 23. PMID 22362038
- [Background] Alter BP, Rosenberg PS, Giri N, Baerlocher GM, Lansdorp PM, Savage SA. Telomere length is associated with disease severity and declines with age in dyskeratosis congenita. Haematologica. 2012 Mar;97(3):353-9. doi: 10.3324/haematol.2011.055269. Epub 2011 Nov 4. PMID 22058220
- [Background] Alter BP, Giri N, Savage SA, Rosenberg PS. Cancer in the National Cancer Institute inherited bone marrow failure syndrome cohort after fifteen years of follow-up. Haematologica. 2018 Jan;103(1):30-39. doi: 10.3324/haematol.2017.178111. Epub 2017 Oct 19. PMID 29051281
- [Derived] Niknafs AM, Giri N, Niewisch MR, Savage SA. Avascular Necrosis and Minimal Trauma Fractures in Telomere Biology Disorders. Clin Genet. 2025 Aug 5. doi: 10.1111/cge.70038. Online ahead of print. PMID 40762130
- [Derived] Raj HA, Lai TP, Niewisch MR, Giri N, Wang Y, Spellman SR, Aviv A, Gadalla SM, Savage SA. The distribution and accumulation of the shortest telomeres in telomere biology disorders. Br J Haematol. 2023 Dec;203(5):820-828. doi: 10.1111/bjh.18945. Epub 2023 Jun 24. PMID 37354000
- [Derived] Bourke G, Wilks D, Kinsey S, Feltbower RG, Giri N, Alter BP. The incidence and spectrum of congenital hand differences in patients with Fanconi anaemia: analysis of 48 patients. J Hand Surg Eur Vol. 2022 Jul;47(7):711-715. doi: 10.1177/17531934221087521. Epub 2022 Mar 31. PMID 35360980
- [Derived] Thompson AS, Giri N, Gianferante DM, Jones K, Savage SA, Alter BP, McReynolds LJ. Shwachman Diamond syndrome: narrow genotypic spectrum and variable clinical features. Pediatr Res. 2022 Dec;92(6):1671-1680. doi: 10.1038/s41390-022-02009-8. Epub 2022 Mar 23. PMID 35322185
- [Derived] Niewisch MR, Giri N, McReynolds LJ, Alsaggaf R, Bhala S, Alter BP, Savage SA. Disease progression and clinical outcomes in telomere biology disorders. Blood. 2022 Mar 24;139(12):1807-1819. doi: 10.1182/blood.2021013523. PMID 34852175
- [Derived] Brodie SA, Khincha PP, Giri N, Bouk AJ, Steinberg M, Dai J, Jessop L, Donovan FX, Chandrasekharappa SC, de Andrade KC, Maric I, Ellis SR, Mirabello L, Alter BP, Savage SA. Pathogenic germline IKZF1 variant alters hematopoietic gene expression profiles. Cold Spring Harb Mol Case Stud. 2021 Aug 2;7(4):a006015. doi: 10.1101/mcs.a006015. Print 2021 Aug. PMID 34162668
- [Derived] Qanash H, Li Y, Smith RH, Linask K, Young-Baird S, Hakami W, Keyvanfar K, Choy JS, Zou J, Larochelle A. Eltrombopag Improves Erythroid Differentiation in a Human Induced Pluripotent Stem Cell Model of Diamond Blackfan Anemia. Cells. 2021 Mar 26;10(4):734. doi: 10.3390/cells10040734. PMID 33810313
- [Derived] Bhar S, Zhou F, Reineke LC, Morris DK, Khincha PP, Giri N, Mirabello L, Bergstrom K, Lemon LD, Williams CL, Toh Y, Elghetany MT, Lloyd RE, Alter BP, Savage SA, Bertuch AA. Expansion of germline RPS20 mutation phenotype to include Diamond-Blackfan anemia. Hum Mutat. 2020 Nov;41(11):1918-1930. doi: 10.1002/humu.24092. Epub 2020 Aug 30. PMID 32790018
- [Derived] Brodie SA, Rodriguez-Aulet JP, Giri N, Dai J, Steinberg M, Waterfall JJ, Roberson D, Ballew BJ, Zhou W, Anzick SL, Jiang Y, Wang Y, Zhu YJ, Meltzer PS, Boland J, Alter BP, Savage SA. 1q21.1 deletion and a rare functional polymorphism in siblings with thrombocytopenia-absent radius-like phenotypes. Cold Spring Harb Mol Case Stud. 2019 Dec 13;5(6):a004564. doi: 10.1101/mcs.a004564. Print 2019 Dec. PMID 31836590
- [Derived] Mirabello L, Khincha PP, Ellis SR, Giri N, Brodie S, Chandrasekharappa SC, Donovan FX, Zhou W, Hicks BD, Boland JF, Yeager M, Jones K, Zhu B, Wang M, Alter BP, Savage SA. Novel and known ribosomal causes of Diamond-Blackfan anaemia identified through comprehensive genomic characterisation. J Med Genet. 2017 Jun;54(6):417-425. doi: 10.1136/jmedgenet-2016-104346. Epub 2017 Mar 9. PMID 28280134
- [Derived] Giri N, Alter BP, Penrose K, Falk RT, Pan Y, Savage SA, Williams M, Kemp TJ, Pinto LA. Immune status of patients with inherited bone marrow failure syndromes. Am J Hematol. 2015 Aug;90(8):702-8. doi: 10.1002/ajh.24046. Epub 2015 May 28. PMID 25963299
- [Derived] Sklavos MM, Stratton P, Giri N, Alter BP, Savage SA, Pinto LA. Reduced serum levels of anti-Mullerian hormone in females with inherited bone marrow failure syndromes. J Clin Endocrinol Metab. 2015 Feb;100(2):E197-203. doi: 10.1210/jc.2014-2838. Epub 2014 Nov 18. PMID 25405500
- [Derived] Alter BP, Giri N, Savage SA, Rosenberg PS. Telomere length in inherited bone marrow failure syndromes. Haematologica. 2015 Jan;100(1):49-54. doi: 10.3324/haematol.2014.114389. Epub 2014 Oct 10. PMID 25304614
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2002-C-0052.html